CLINICAL TRIAL: NCT05618262
Title: Evaluation of the Emergency Imaging Strategy for the Diagnostic Management of Renal Colic
Acronym: Renal-Colic
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7634
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Renal Colic
Keywords: Renal Colic; Nephritic Colic; Pyelocalic dilatation
MeSH Terms: conditions — Renal Colic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emergency imaging is necessary for the diagnostic management of renal colic in the emergency department. Ultrasound is rapidly available and non-irradiating, allowing to look for a stone and a pyelocalic dilatation. But it is less sensitive when the stone is ureteral. CT has a sensitivity of 96% and a specificity of 100%. The latest French recommendations date from 2008, recommending ultrasound and an unprepared abdomen in cases of uncomplicated renal colic. For the European Society of Radiology, ultrasound should be the first-line examination. The place of a systematic CT scan as first-line examination for the diagnosis of renal colic in the emergency department is therefore still under discussion.

An evaluation of practice will make it possible to assess the imaging strategy applied in an emergency department.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years)
* Subject who was managed in the NHC emergency department from July 01, 2018 to June 30, 2019 with a final diagnosis of renal colic diagnostic
* Subject who has not expressed opposition, after information, to the reuse of their data for the purpose of this research

Exclusion criteria:

* Subject who has expressed opposition to participating in the study
* Subject under guardianship or curatorship
* Subject under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years) who was managed in the NHC emergency department from July 01, 2018 to June 30, 2019 with a final diagnosis of renal colic diagnostic
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Retrospective study of the practices of management of renal colic in the emergency room concerning the imaging strategy | Files analysed retrospectively from from July 01, 2018 to June 30, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'accueil des urgences - CHU de Strasbourg - France, Strasbourg, France